CLINICAL TRIAL: NCT02746796
Title: ONO-4538 Phase II/III Study A Multicenter, Randomized Study in Patients With Unresectable Advanced or Recurrent Gastric Cancer
Brief Title: Study of ONO-4538 in Gastric Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-4538-37
Record Dates: First submitted 2016-03-29; First posted 2016-04-21 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ONO-4538 + SOX Therapy Cohort (Part 1) (Experimental): ONO-4538 360 mg solution intravenously for 30 min in every 3 weeks. Oxaliplatin 130 mg/m2 (BSA) solution intravenously for 2 hours once-daily, followed by 20 days off.
  Tegafur-gimeracil-oteracil potassium combination drug 40 - 60 mg bid orally in 14 days, followed by 7 days off Each drug will be continued until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
  Interventions: Drug: ONO-4538; Drug: Oxaliplatin; Drug: Tegafur- Gimeracil-Oteracil potassium
- ONO-4538 + CapeOX Therapy Cohort (Part 1) (Experimental): ONO-4538 360 mg solution intravenously for 30 min in every 3 weeks. Oxaliplatin 130 mg/m2 (body surface area) solution intravenously for 2 hours once-daily, followed by 20 days off.
  Capecitabine 1200 - 2100 mg bid orally in 14 days, followed by 7 days off. Each drug will be continued until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
  Interventions: Drug: ONO-4538; Drug: Oxaliplatin; Drug: Capecitabine
- ONO-4538 + chemotherapy group (Part 2) (Experimental): With regard to the ONO-4538 + chemotherapy group, either SOX therapy or CapeOX therapy will be selected as the chemotherapy by the investigator or the subinvestigator, taking into account the condition of each subject.
  ONO-4538 360 mg solution intravenously for 30 min in every 3 weeks. Oxaliplatin 130 mg/m2 (body surface area) solution intravenously for 2 hours once-daily, followed by 20 days off.
  Tegafur-gimeracil-oteracil potassium combination drug 40 - 60 mg bid or Capecitabine 1000 mg/ m2 (body surface area) bid orally in 14 days, followed by 7 days off.
  Each drug will be continued until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
  Interventions: Drug: ONO-4538; Drug: Oxaliplatin; Drug: Tegafur- Gimeracil-Oteracil potassium; Drug: Capecitabine
- Placebo + Chemotherapy group (Part 2) (Placebo Comparator): With regard to the placebo + chemotherapy group, either SOX therapy or CapeOX therapy will be selected as the chemotherapy by the investigator or the subinvestigator, taking into account the condition of each subject.
  Placebo solution intravenously for 30 min in every 3 weeks. Oxaliplatin 130 mg/m2 (body surface area) solution intravenously for 2 hours once-daily, followed by 20 days off.
  Tegafur-gimeracil-oteracil potassium combination drug 40 - 60 mg bid or Capecitabine 1000 mg/ m2 (body surface area) bid orally in 14 days, followed by 7 days off.
  Each drug will be continued until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
  Interventions: Drug: Oxaliplatin; Drug: Tegafur- Gimeracil-Oteracil potassium; Drug: Capecitabine; Drug: Placebo

INTERVENTIONS:
Drug: ONO-4538
  Arms: ONO-4538 + CapeOX Therapy Cohort (Part 1); ONO-4538 + SOX Therapy Cohort (Part 1); ONO-4538 + chemotherapy group (Part 2)
Drug: Oxaliplatin
Drug: Tegafur- Gimeracil-Oteracil potassium
  Arms: ONO-4538 + SOX Therapy Cohort (Part 1); ONO-4538 + chemotherapy group (Part 2); Placebo + Chemotherapy group (Part 2)
Drug: Capecitabine
  Arms: ONO-4538 + CapeOX Therapy Cohort (Part 1); ONO-4538 + chemotherapy group (Part 2); Placebo + Chemotherapy group (Part 2)
Drug: Placebo
  Arms: Placebo + Chemotherapy group (Part 2)

SUMMARY:
The purpose of study is to evaluate the efficacy and safety of ONO-4538 with chemotherapy in unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer) not previously treated with the first-line therapy. Part 1 is intended to evaluate the tolerability, safety, and efficacy of ONO-4538 in combination with SOX therapy (Tegafur / gimeracil / oteracil potassium + Oxaliplatin) or CapeOX therapy (Capecitabine + Oxaliplatin). In part 2, the investigator or the subinvestigator will choose a chemotherapy (SOX or CapeOX therapy), taking into account the condition of each subject. Part 2 is planned to evaluate the efficacy and safety of ONO-4538 + chemotherapy in comparison with placebo + chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer) that has not been treated with the first-line therapy with systemic antitumor agents for advanced or recurrent gastric cancer (including esophagogastric junction cancer)
* Have measurable lesions as defined in RECIST Guideline Version 1.1
* ECOG PS score 0 or 1
* Have a life expectancy of at least 3 months

Exclusion Criteria:

* Have multiple cancers
* Have a current or past history of severe hypersensitivity to any other antibody products
* Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment
* Patients with active, known or suspected autoimmune disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (central assessment by IRRC) (only Part 2) | Up to study completion (estimated time frame: 48 months)
Overall survival (only Part 2) | Up to study completion (estimated time frame: 54 months)

SECONDARY OUTCOMES:
Objective response rate (only Part 2) | Up to study completion (estimated time frame: 54 months)
Progression-free survival (assessment by the site investigator)(only Part 2) | Up to study completion (estimated time frame: 54 months)
Duration of response (only Part 2) | Up to study completion (estimated time frame: 54 months)
Disease control rate (only Part 2) | Up to study completion (estimated time frame: 54 months)
Time to response (only Part 2) | Up to study completion (estimated time frame: 54 months)
Best overall response (only Part 2) | Up to study completion (estimated time frame: 54 months)
Percent change in the sum of diameters of target lesions (only Part 2) | Up to study completion (estimated time frame: 54 months)
Safety will be analyzed through the incidence of adverse events, serious adverse events | Up to 28 days from last dose
Safety will be analyzed through the incidence of laboratory abnormalities | Up to 28 days from last dose

CONTACTS AND LOCATIONS:
Overall Officials: Mitsunobu Tanimoto, Study Director — Ono Pharmaceutical Co. Ltd
Locations (130):
- Japan (97):
  - Aichi Clinical Site, Nagoya, Aichi-ken
  - Aomori Clinical Site, Hirosaki, Aomori
  - Aomori Clinical Site, Misawa, Aomori
  - Chiba Clinical Site, Funabashi, Chiba
  - Chiba Clinical Site, Kamogawa, Chiba
  - Chiba Clinical Site, Kashiwa, Chiba
  - Ehime Clinical Site1, Matsuyama, Ehime
  - Ehime Clinical Site2, Matsuyama, Ehime
  - Fukuoka Clinical Site, Iizuka, Fukuoka
  - Fukuoka Clinical Site1, Kitakyushu, Fukuoka
  - Fukuoka Clinical Site2, Kitakyushu, Fukuoka
  - Fukuoka Clinical Site, Kurume, Fukuoka
  - Gifu Clinical Site, Gifu, Gifu
  - Gifu Clinical Site, Ōgaki, Gifu
  - Gumma Clinical Site, Maebashi, Gunma
  - Gunma Clinical Site, Ōta, Gunma
  - Gumma Clinical Site, Takasaki, Gunma
  - Hiroshima Clinical Site, Kure, Hiroshima
  - Hokkaido Clinical Site, Hakodate, Hokkaido
  - Hokkaido Clinical Site1, Sapporo, Hokkaido
  - Hokkaido Clinical Site2, Sapporo, Hokkaido
  - Hokkaido Clinical Site3, Sapporo, Hokkaido
  - Hokkaido Clinical Site4, Sapporo, Hokkaido
  - Hyogo Clinical Site, Akashi, Hyōgo
  - Hyogo Clinical Site, Amagasaki, Hyōgo
  - Hyogo Clinical Site, Kobe, Hyōgo
  - Hyogo Clinical Site, Nishinomiya, Hyōgo
  - Ibaraki Clinical Site, Higashiibaraki-gun, Ibaraki
  - Ibaraki Clinical Site, Tsuchiura-shi, Ibaraki
  - Ishikawa Clinical Site1, Kanazawa, Ishikawa-ken
  - Ishikawa Clinical Site2, Kanazawa, Ishikawa-ken
  - Iwate Clinical Site, Morioka, Iwate
  - Kagawa Clinical Site, Kita-gun, Kagawa-ken
  - Kanagawa Clinical Site, Isehara, Kanagawa
  - Kanagawa Clinical Site, Kamakura, Kanagawa
  - Kanagawa Clinical Site, Sagamihara, Kanagawa
  - Kanagawa Clinical Site1, Yokohama, Kanagawa
  - Kanagawa Clinical Site2, Yokohama, Kanagawa
  - Kanagawa Clinical Site3, Yokohama, Kanagawa
  - Miyagi Clinical Site, Natori-shi, Miyagi
  - Miyagi Clinical Site, Ōsaki, Miyagi
  - Miyagi Clinical Site, Sendai, Miyagi
  - Nagano Clinical Site, Saku, Nagano
  - Nara Clinical Site, Ikoma, Nara
  - Nara Clinical Site, Kashihara-shi, Nara
  - Okayama Clinical Site, Kurashiki, Okayama-ken
  - Osaka Clinical Site, Izumi, Osaka
  - Osaka Clinical Site, Sakai, Osaka
  - Osaka Clinical Site, Sayama, Osaka
  - Osaka Clinical Site, Suita, Osaka
  - Osaka Clinical Site, Takatsuki, Osaka
  - Osaka Clinical Site, Toyonaka, Osaka
  - Saitama Clinical Site, Hidaka, Saitama
  - Saitama Clinical Site, Kitaadachi-gun, Saitama
  - Shizuoka Clinical Site, Hamamatsu, Shizuoka
  - Tochigi Clinical Site, Shimotsuke, Tochigi
  - Tochigi Clinical Site, Utsunomiya, Tochigi
  - Tokyo Clinical Site, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site, Chuo-ku, Tokyo
  - Tokyo Clinical Site, Fuchū, Tokyo
  - Tokyo Clinical Site, Koto-ku, Tokyo
  - Tokyo Clinical Site, Minato-ku, Tokyo
  - Tokyo Clinical Site, Shinagawa-ku, Tokyo
  - Tokyo Clinical Site1, Shinjuku-ku, Tokyo
  - Tokyo Clinical Site2, Shinjuku-ku, Tokyo
  - Tokyo Clinical Site, Tachikawa, Tokyo
  - Tottori Clinical Site, Yonago, Tottori
  - Yamagata Clinical Site, Sakata, Yamagata
  - Akita Clinical Site, Akita
  - Chiba Clinical Site1, Chiba
  - Chiba Clinical Site2, Chiba
  - Fukui Clinical Site, Fukui
  - Fukuoka Clinical Site1, Fukuoka
  - Fukuoka Clinical Site2, Fukuoka
  - Fukuoka Clinical Site3, Fukuoka
  - Fukuoka Clinical Site4, Fukuoka
  - Fukushima Clinical Site, Fukushima
  - Hiroshima Clinical Site1, Hiroshima
  - Hiroshima Clinical Site2, Hiroshima
  - Hiroshima Clinical Site3, Hiroshima
  - Kumamoto Clinical Site1, Kumamoto
  - Kumamoto Clinical Site2, Kumamoto
  - Kumamoto Clinical Site3, Kumamoto
  - Kyoto Clinical Site1, Kyoto
  - Kyoto Clinical Site2, Kyoto
  - Kyoto Clinical Site3, Kyoto
  - Niigata Clinical Site, Niigata
  - Okayama Clinical Site, Okayama
  - Osaka Clinical Site1, Osaka
  - Osaka Clinical Site2, Osaka
  - Osaka Clinical Site3, Osaka
  - Osaka Clinical Site4, Osaka
  - Shizuoka Clinical Site, Shizuoka
  - Tokushima Clinical Site, Tokushima
  - Toyama Clinical Site, Toyama
  - Wakayama Clinical Site, Wakayama
  - Yamagata Clinical Site, Yamagata
- South Korea (23):
  - Gyeongnam Clinical Site, Gyeongnam, Gyeongsangnam-do
  - Busan Clinical Site, Busan
  - Daegu Clinical Site 1, Daegu
  - Daegu Clinical Site 2, Daegu
  - Daejeon Clinical Site, Daejeon
  - Gyeonggi-Do Clinical Site1, Gyeonggi-do
  - Gyeonggi-Do Clinical Site2, Gyeonggi-do
  - Gyeonggi-Do Clinical Site3, Gyeonggi-do
  - Gyeonggi-Do Clinical Site4, Gyeonggi-do
  - Gyeonggi-Do Clinical Site5, Gyeonggi-do
  - Incheon Clinical Site, Incheon
  - Jeollabuk-Do Clinical Site, Jeollabuk-Do
  - Jeollanam-do Clinical Site, Jeollanam-do
  - Seoul Clinical Site 1, Seoul
  - Seoul Clinical Site 2, Seoul
  - Seoul Clinical Site 3, Seoul
  - Seoul Clinical Site 4, Seoul
  - Seoul Clinical Site 5, Seoul
  - Seoul Clinical Site 6, Seoul
  - Seoul Clinical Site7, Seoul
  - Seoul Clinical Site8, Seoul
  - Seoul Clinical Site9, Seoul
  - Ulsan Clinical Site, Ulsan
- Taiwan (10):
  - Kaohsiung Clinical Site1, Kaohsiung City
  - Kaohsiung Clinical Site2, Kaohsiung City
  - New Taipei Clinical Site 1, New Taipei City
  - Taichung Clinical Site 1, Taichung
  - Taichung Clinical Site2, Taichung
  - Tainan Clinical Site1, Tainan
  - Tainan Clinical Site2, Tainan
  - Taipei Clinical Site1, Taipei
  - Taipei Clinical Site2, Taipei
  - Taoyuan Clinical Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boku N, Omori T, Shitara K, Sakuramoto S, Yamaguchi K, Kato K, Kadowaki S, Tsuji K, Ryu MH, Oh DY, Oh SC, Rha SY, Lee KW, Chung IJ, Sym SJ, Chen LT, Chen JS, Bai LY, Nakada T, Hagihara S, Makino R, Nishiyama E, Kang YK. Nivolumab plus chemotherapy in patients with HER2-negative, previously untreated, unresectable, advanced, or recurrent gastric/gastroesophageal junction cancer: 3-year follow-up of the ATTRACTION-4 randomized, double-blind, placebo-controlled, phase 3 trial. Gastric Cancer. 2024 Nov;27(6):1287-1301. doi: 10.1007/s10120-024-01535-0. Epub 2024 Aug 20. PMID 39162872
- [Derived] Kang YK, Chen LT, Ryu MH, Oh DY, Oh SC, Chung HC, Lee KW, Omori T, Shitara K, Sakuramoto S, Chung IJ, Yamaguchi K, Kato K, Sym SJ, Kadowaki S, Tsuji K, Chen JS, Bai LY, Oh SY, Choda Y, Yasui H, Takeuchi K, Hirashima Y, Hagihara S, Boku N. Nivolumab plus chemotherapy versus placebo plus chemotherapy in patients with HER2-negative, untreated, unresectable advanced or recurrent gastric or gastro-oesophageal junction cancer (ATTRACTION-4): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):234-247. doi: 10.1016/S1470-2045(21)00692-6. Epub 2022 Jan 11. PMID 35030335
- [Derived] Boku N, Ryu MH, Kato K, Chung HC, Minashi K, Lee KW, Cho H, Kang WK, Komatsu Y, Tsuda M, Yamaguchi K, Hara H, Fumita S, Azuma M, Chen LT, Kang YK. Safety and efficacy of nivolumab in combination with S-1/capecitabine plus oxaliplatin in patients with previously untreated, unresectable, advanced, or recurrent gastric/gastroesophageal junction cancer: interim results of a randomized, phase II trial (ATTRACTION-4). Ann Oncol. 2019 Feb 1;30(2):250-258. doi: 10.1093/annonc/mdy540. PMID 30566590